CLINICAL TRIAL: NCT03913325
Title: Early Identification of Risk for and Prevention of Sickness Absence Due to Musculoskeletal Pain (PREVSAM) - a Randomized Controlled Trial
Brief Title: Early Identification of Risk for and Prevention of Sickness Absence Due to Musculoskeletal Pain - an RCT
Acronym: PREVSAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Swedish Council for Working Life and Social Research (Other)
Responsible Party: Principal Investigator, Maria Larsson, Associate Professor, Vastra Gotaland Region
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FORTE 2018-01250
Record Dates: First submitted 2019-04-09; First posted 2019-04-12 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Musculoskeletal Disorder
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PREVSAM model (Experimental)
  Interventions: Other: PREVSAM model
- Treatment as usual (Active Comparator)
  Interventions: Other: Treatment as usual (standard treatment)

INTERVENTIONS:
Other: PREVSAM model — A person-centred rehabilitation plan, including coordinated measures within primary health care as well as in collaboration with participants' employers, and when relevant the Swedish Public Employment Agency
  Arms: PREVSAM model
Other: Treatment as usual (standard treatment) — Treatment as usual (ordinary/standard) treatment. Can include unimodal or multimodal treatment of physiotherapy solely and/or occupational therapy
  Arms: Treatment as usual

SUMMARY:
Background: Musculoskeletal pain is a leading cause of disability in the world. Although the majority of musculoskeletal-related pain conditions, such as low back pain, often resolves spontaneously, pain may recur or persist over a long time, potentially leading to disability and subsequent reduced work capacity and long-term sickness absence. There is a need for early identification of individuals in which this may occur, to prevent or reduce the risk of long-term musculoskeletal pain and long-term sickness absence. The aim of the trial described in this protocol is to evaluate a primary care rehabilitation model, PREVSAM, including early identification of patients at risk for long-term musculoskeletal pain and related sickness absence and a coordinated interdisciplinary rehabilitation programme based on individual and organizational resources.

Methods: Eligible individuals will be recruited from primary care rehabilitation centres, health care centres, and include those who seek care for musculoskeletal pain and who are at risk of developing persistent pain, disability and sickness absence. Participants will be randomized to either treatment according to the PREVSAM model (intervention group) or treatment as usual (TAU) within primary care (control group). The PREVSAM model will comprise a person-centred rehabilitation plan, including coordinated measures within primary health care as well as in collaboration with participants' employers, and when relevant the Swedish Public Employment Agency. The primary outcome sickness absence will be measured at 3 and12 months from the Swedish Social Insurance Agency regarding: the number and proportion of individuals who remain in full- or part-time work, the number of gross and net days of sickness during the follow-up period, and time to first sickness absence spell. Secondary outcomes are patient-reported work ability, pain, health-related quality of life, risk for sickness absence, anxiety/depression, general and pain self-efficacy and disability at 3 months after inclusion (short-term follow-up), and at 6 and 12 months (long-term follow-up). Follow-up of drug consumption and cost-effectiveness analyes will be performed at 12 months.

Discussion: This study is expected to provide new knowledge on how to best identify individuals at risk for long-term disability and sick leave due to musculoskeletal pain, and whether rehabilitation according to the PREVSAM model is effective. The study findings may contribute to more effective primary care rehabilitation processes of this large patient population, and potentially reduce sick leave and costs for healthcare and society.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18
* Musculoskeletal pain, preferably less than 3 months
* Risk for development of persistent musculoskeletal pain and disability ≥ 40 p on ÖMPSQ-SF
* Independently mobile (with or without aids), to be capable of participating in intervention

Exclusion Criteria:

* Pain not primarily generated from the musculoskeletal system
* Sickness cash benefit more than 30 days during the last 12 months due to pain from the musculoskeletal system
* Full disability pension
* Pregnancy
* Red flag disorders such as malignancy/cancer, acute traumas such as fracture (less than 6 months ago) or infection, spinal cord compression/cauda equina
* Severe mental illness

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Registered sickness absence | During 12 months from baseline
  Registered sickness absence at Swedish Social Insurance Agency

SECONDARY OUTCOMES:
Short time sickness absence | Weekly for 12 months following baseline
  Self reported sickness absence by text messages
Patient reported work ability | At 1, 3, 6 and 12 months following baseline
  Self reported work ability using single question of Work Ability Index (WAI) (NRS 0-10)
Risk of sickness absence assessed by Örebro Musculoskeletal Pain Screening Questionnaire Short Form (ÖMPSQ-SF) | At 1, 3, 6 and 12 months following baseline
  Self reported risk of sickness absence using ÖMPSQ (NRS 0-10)
Patient reported pain duration | At 1, 3, 6 and 12 months following baseline
  Self reported pain duration
Patient reported pain intensity | At 1, 3, 6 and 12 months following baseline
  Self reported pain intensity
Patient reported pain widespread | At 1, 3, 6 and 12 months following baseline
  Self reported pain widespread
Health Related Quality of Life (HRQL) assessed by EuroQol 5 dimensions | At 1, 3, 6 and 12 months following baseline
  Self reported HRQL using EQ5D (5 dimensions with 3 answering options which form an index)
Health Related Quality of Life (HRQL) assessed by EuroQol VAS (0-100) | At 1, 3, 6 and 12 months following baseline
  Self reported HRQL using EQVAS
Anxiety and Depression assessed by Hospital Anxiety and Depression Scale (HADS) | At 1, 3, 6 and 12 months following baseline
  Self reported anxiety and depression using HADS (NRS 0-21 per Anxiety and depression respectively)
Function/Disability assessed by Disability Rating Index (DRI) | At 1, 3, 6 and 12 months following baseline
  Self reported function/disability assessed by Disability Rating Index (DRI) (10 VAS summed range 0-100)
Drug use | 3 months before to 12 months after baseline
  Use of drugs/medication collected from "Läkemedelsregistret"
General self-efficacy | At 1, 3, 6 and 12 months following baseline
  Self reported general self efficacy assessed by General self-efficacy scale; the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Pain Self-efficacy scale 2 items | At 1, 3, 6 and 12 months following baseline
  Self reported pain self efficacy assessed by PSEQ-2SV; the total score ranges between 0 and 12, with a higher score indicating more pain self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Research and Development primary care Region Västra Götaland, Gothenburg, Västra Götalandregionen, Sweden

REFERENCES:
- [Derived] Larsson M, Nordeman L, Holmgren K, Grimby-Ekman A, Hensing G, Bjorkelund C, Bergman S, Ekhammar A, Dottori M, Bernhardsson S. Prevention of sickness absence through early identification and rehabilitation of at-risk patients with musculoskeletal pain (PREVSAM): a randomised controlled trial protocol. BMC Musculoskelet Disord. 2020 Nov 28;21(1):790. doi: 10.1186/s12891-020-03790-5. PMID 33248457